CLINICAL TRIAL: NCT00953732
Title: A 12 Month, Long-term Follow-up Study of Patients With Actinic Keratosis on the Head (Face or Scalp) Who Have Completed Day 57 in Studies PEP005-016 or PEP005-025 (REGION IIa and IIb)
Brief Title: A Long Term Follow up Study of Patients Who Have Completed the PEP005-016 or PEP005-025 Studies
Status: Completed | Type: Observational
Sponsor: Peplin (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP005-030
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Actinic Keratosis
Keywords: Peplin; Actinic keratosis; PEP005
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Lesion count

INTERVENTIONS:
Drug: Lesion count — Lesion count in area treated by study drug in a prior study. No drug will be applied during this long-term follow up study. Drug was applied during the primary study.
  Other Names: AK lesion recurrence

SUMMARY:
This study is designed to follow up patients who have achieved complete clearance of AK lesions at the Day 57 visit having completed the PEP005-016 or PEP005-025 studies over a 12 month period to assess both recurrence of Actinic Keratosis (AK) lesions and long term safety in the selected treatment area.

DETAILED DESCRIPTION:
A 12 month long-term follow-up study of patients who have achieved complete clearance of AK lesions at the Day 57 in the Phase 3 studies PEP005-016 or PEP005-025.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have achieved complete clearance of AK lesions (lesion count = 0) at Day 57 in one of the following Peplin AK clinical studies: PEP005-016 or PEP005-025
* Patient has provided informed consent documented by signing the Informed Consent Form (ICF) prior to any study-related procedures

Exclusion Criteria:

* Concurrent participation in another research study which would involve the selected treatment area (except for any post-study follow-up visits for previous Peplin AK study)
* Early termination from study PEP005-016 or PEP005-025

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients must have achieved complete clearance of AK lesions at Day 57 visit in either study PEP005-016 or PEP005-025 will be offered participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Summarize treatment area recurrence of AK lesions, in the selected treatment area | 12 months

SECONDARY OUTCOMES:
Summarize long-term safety data(incidence of AEs in the treatment area) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Bauer, MD, Study Director — Chief Medical Officer
Locations (42):
- United States (38):
  - Burke Pharmaceutical Research, Hot Springs, Arizona
  - Center for Dermatology, Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Dermatology Specialists Inc, Oceanside, California
  - Skin Surgery Medical Group Inc., San Diego, California
  - Conant Medical Group, San Francisco, California
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - University of Miami, Skin Research Camp, Miami, Florida
  - Atlanta Dermatology, Vein & Research Center, LLC, Alpharetta, Georgia
  - Medaphase Inc, Newnan, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Glazer Dermatology, Buffalo Grove, Illinois
  - Laser Skin Surgery Center of Indiana, Carmel, Indiana
  - Deaconess Clinic, Inc, Evansville, Indiana
  - Dawes Fretein Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Pedia Research LLC, Owensboro, Kentucky
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialists, PC, Omaha, Nebraska
  - Karl G. Heine Dermatology, Henderson, Nevada
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - Dermatology Associates of Rochester, PC, Rochester, New York
  - Dermatology, Laser Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Oregon Medical Research, Portland, Oregon
  - Dermatology Research Associates, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - J & S Studies, Inc., College Station, Texas
  - Suzanne Bruce and Associates, The Center for Skin Research, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Dermatology Associates of Tyler, Tyler, Texas
  - Center for Clinical Studies, Webster, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - The Education and Research Foundation, Lynchburg, Virginia
  - Virginia Clinical Research, Inc, Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington
- Australia (4):
  - Southderm Pty Ltd, Kogarah, New South Wales
  - St George Dematology and Skin Cancer Centre, Kogarah, New South Wales
  - The Skin Centre, Benowa, Queensland
  - South East Dermatology, Belmont Specialist Centre, Carina Heights, Queensland

REFERENCES:
- [Derived] Lebwohl M, Shumack S, Stein Gold L, Melgaard A, Larsson T, Tyring SK. Long-term follow-up study of ingenol mebutate gel for the treatment of actinic keratoses. JAMA Dermatol. 2013 Jun;149(6):666-70. doi: 10.1001/jamadermatol.2013.2766. PMID 23553119
- See also: Food and Drug Authority — http://www.fda.gov
- See also: Therapeutic Goods Administration — http://www.tga.gov.au